CLINICAL TRIAL: NCT06522971
Title: Exploration of the Molecular Mechanisms Behind the Effects of Physical Exercise on Response to Neoadjuvant Chemotherapy in Breast Cancer Patients
Brief Title: Effects of Physical Exercise on Response to Treatement in Breast Cancer
Acronym: CancerBeat
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Latvian Biomedical Research and Study Centre (Other Government)
Collaborators: Riga East Clinical University Hospital (Other Government); Latvian Academy of Sport Education (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: NFI_164
Record Dates: First submitted 2024-07-09; First posted 2024-07-26 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: High intensity interval training
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-intensity interval training (HIIT) (Experimental): High-intensity interval training during neoadjuvant chemotherapy
  Interventions: Behavioral: High-intensiy interval training
- Low level of physical activity (CON) (No Intervention): Advised to maintain usual level of physical activity during neoadjuvant chemotherapy

INTERVENTIONS:
Behavioral: High-intensiy interval training — All participants undergo physical capacity tests before the onset of NAC and after the last course of NAC but before the breast cancer surgery. A treadmill protocol consisting of twenty-one 1-minute stages, with speed and/or grade increments at each stage, is used to obtain VO2 peak (the highest amount of oxygen consumed at peak exercise) data. The HIIT intervention consists of 2 to 3 exercise sessions per week for 6 months. The HIIT session starts with a 6-minute warm-up period at about 65-70% of maximal heart rate (HRmax) followed by 4 X 4-min high-intensity intervals (85%-95% of HRmax) combined with 3 min period of active recovery (55-70% of HRmax).
  Arms: High-intensity interval training (HIIT)

SUMMARY:
The goal of this clinical trial is to learn how regular physical exercise affects breast cancer patients' response to standard neoadjuvant chemotherapy (NAC) and to gain an insight into the molecular mechanisms underlying the effects of exercise on cancer biology. of exercise-induced alterations in cancer gene expression and the immune tumor microenvironment. The main questions it aims to answer are:

* Does a high-intensity interval training (HIIT) program during treatment improve patients' response to NAC and quality of life as compared to low level of physical activity during the treatment?
* What are the differences in the residual tumor gene expression and tumor infiltrating immune cell profile between patients taking HIIT during the NAC and patients with low level of physical activity?
* What are the roles of extracellular vesicles (EVs) in mediating the effects of exercise on cancer progression?

Patients in HIIT group will undergo a personalized HIIT program consisting of 3 training sessions per week for the whole duration of NAC, whereas patients from the control group (Ctrl) will be advised to maintain their usual level of physical activity during NAC. After the breast surgery, response to NAC will be assessed by Miller-Payne grading. Tumor and normal breast tissue specimens will be collected for RNA sequencing analysis. Blood samples will be collected before and immediately after the training for the analysis of RNA and protein cargo of circulating EVs.

ELIGIBILITY:
Inclusion criteria:

* Primary breast cancer; stage IIA-B, IIIA-C (TNM: T1-4, N0-3, M0) at diagnosis
* Diagnosis established by core needle biopsy
* Age 30-65 years
* Prescribed doxorubicin/cyclophosphamide-based NAC
* Oral and written consent

Exclusion criteria:

* Cardiac pathologies
* Pregnancy
* Blood transfusion in the last six months
* Another oncological disease
* Previous chemotherapy, hormonal or X-ray treatment
* Participation in another clinical trial
* Currently performing more than 180 min of moderate to high intensity aerobic training per week

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Miller-Payne grade | 6 months
  Response to NAC assessed by histological examination of residual tumor at surgery using Miller-Payne grading from 1 to 5, where grade 1 means no response or some alterations to individual malignant cells but no reduction in overall cellularity, whereas grade 5 is a pathological complete response.
Gene expression profile | 12 months
  Alterations in the tumor gene expression profile will be assessed by RNA sequencing of surgical tumor and normal breast tissue specimens

SECONDARY OUTCOMES:
RNA cargo of extracellular vesicles | Before intervention and after 6 months
  Exercise-induced alterations in the RNA cargo of circulating extracellular vesicles will be studied by RNA sequencing
Protein cargo of extracellular vesicles | Before intervention and after 6 months
  Exercise-induced alterations in the protein cargo of circulating extracellular vesicles will be studied by proteomic analysis
Number and phenotype of tumor-infiltrating immune cells | 12 months
  Immunophenotyping of tumor-infiltrating immune cells will be performed by multiplex immunofluorescence in breast tumor tissue specimens
Global health-related quality of life | 6 months
  Global health-related quality of life will be assessed by the European Organisation for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30). All scales and single-item measures yield scores ranging from 0 to 100. A high score on a functional scale indicates superior functioning and a high score on the global health status/QoL scale indicates a high quality of life. Conversely, a high score on a symptom scale or item indicates a heightened level of health complaints and/ or presence of treatment side effects.
Breast cancer-related quality of life | 6 months
  Breast cancer-related quality of life assessed by the European Organisation for Research and Treatment of Cancer Breast cancer module (EORTC QLQ-B23) questionnaire that includes 23 questions addressing disease symptoms, treatment side effects, body image, sexual functioning, and future perspectives. All scales and single-item measures yield scores ranging from 0 to 100.
VO2 peak | Before intervention and after 6 months
  Oxygen peak consumption will be measured by UNCCRI treadmill protocol
30 sec sit-to-stand test | Before intervention and after 6 months
  The number of sit- and stand-up movement repetitions achieved during 30 sec will be recorded
6-minute walk test | Before intervention and after 6 months
  The test will be performed indoors on 30 m long testing course and length of walked distance will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Aija Linē, PhD, Principal Investigator — Latvian Biomedical Research and Study Centre
Locations (1):
- Latvian Biomedical Research and Study centre, Riga, Select One, Latvia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moore SC, Lee IM, Weiderpass E, Campbell PT, Sampson JN, Kitahara CM, Keadle SK, Arem H, Berrington de Gonzalez A, Hartge P, Adami HO, Blair CK, Borch KB, Boyd E, Check DP, Fournier A, Freedman ND, Gunter M, Johannson M, Khaw KT, Linet MS, Orsini N, Park Y, Riboli E, Robien K, Schairer C, Sesso H, Spriggs M, Van Dusen R, Wolk A, Matthews CE, Patel AV. Association of Leisure-Time Physical Activity With Risk of 26 Types of Cancer in 1.44 Million Adults. JAMA Intern Med. 2016 Jun 1;176(6):816-25. doi: 10.1001/jamainternmed.2016.1548. PMID 27183032
- [Background] Matthews CE, Moore SC, Arem H, Cook MB, Trabert B, Hakansson N, Larsson SC, Wolk A, Gapstur SM, Lynch BM, Milne RL, Freedman ND, Huang WY, Berrington de Gonzalez A, Kitahara CM, Linet MS, Shiroma EJ, Sandin S, Patel AV, Lee IM. Amount and Intensity of Leisure-Time Physical Activity and Lower Cancer Risk. J Clin Oncol. 2020 Mar 1;38(7):686-697. doi: 10.1200/JCO.19.02407. Epub 2019 Dec 26. PMID 31877085
- [Background] Hornsby WE, Douglas PS, West MJ, Kenjale AA, Lane AR, Schwitzer ER, Ray KA, Herndon JE 2nd, Coan A, Gutierrez A, Hornsby KP, Hamilton E, Wilke LG, Kimmick GG, Peppercorn JM, Jones LW. Safety and efficacy of aerobic training in operable breast cancer patients receiving neoadjuvant chemotherapy: a phase II randomized trial. Acta Oncol. 2014 Jan;53(1):65-74. doi: 10.3109/0284186X.2013.781673. Epub 2013 Aug 19. PMID 23957716
- [Background] Mijwel S, Backman M, Bolam KA, Olofsson E, Norrbom J, Bergh J, Sundberg CJ, Wengstrom Y, Rundqvist H. Highly favorable physiological responses to concurrent resistance and high-intensity interval training during chemotherapy: the OptiTrain breast cancer trial. Breast Cancer Res Treat. 2018 May;169(1):93-103. doi: 10.1007/s10549-018-4663-8. Epub 2018 Jan 18. PMID 29349712
- [Background] Li Y, Xiao X, Zhang Y, Tang W, Zhong D, Liu T, Zhu Y, Li J, Jin R. Effect of Exercise on Breast Cancer: A Systematic Review and Meta-analysis of Animal Experiments. Front Mol Biosci. 2022 Jun 6;9:843810. doi: 10.3389/fmolb.2022.843810. eCollection 2022. PMID 35733941
- [Background] Hagar A, Wang Z, Koyama S, Serrano JA, Melo L, Vargas S, Carpenter R, Foley J. Endurance training slows breast tumor growth in mice by suppressing Treg cells recruitment to tumors. BMC Cancer. 2019 Jun 4;19(1):536. doi: 10.1186/s12885-019-5745-7. PMID 31164094
- [Background] Wennerberg E, Lhuillier C, Rybstein MD, Dannenberg K, Rudqvist NP, Koelwyn GJ, Jones LW, Demaria S. Exercise reduces immune suppression and breast cancer progression in a preclinical model. Oncotarget. 2020 Jan 28;11(4):452-461. doi: 10.18632/oncotarget.27464. eCollection 2020 Jan 28. PMID 32064049
- [Background] Pedersen L, Idorn M, Olofsson GH, Lauenborg B, Nookaew I, Hansen RH, Johannesen HH, Becker JC, Pedersen KS, Dethlefsen C, Nielsen J, Gehl J, Pedersen BK, Thor Straten P, Hojman P. Voluntary Running Suppresses Tumor Growth through Epinephrine- and IL-6-Dependent NK Cell Mobilization and Redistribution. Cell Metab. 2016 Mar 8;23(3):554-62. doi: 10.1016/j.cmet.2016.01.011. Epub 2016 Feb 16. PMID 26895752
- [Background] Yanez-Mo M, Siljander PR, Andreu Z, Zavec AB, Borras FE, Buzas EI, Buzas K, Casal E, Cappello F, Carvalho J, Colas E, Cordeiro-da Silva A, Fais S, Falcon-Perez JM, Ghobrial IM, Giebel B, Gimona M, Graner M, Gursel I, Gursel M, Heegaard NH, Hendrix A, Kierulf P, Kokubun K, Kosanovic M, Kralj-Iglic V, Kramer-Albers EM, Laitinen S, Lasser C, Lener T, Ligeti E, Line A, Lipps G, Llorente A, Lotvall J, Mancek-Keber M, Marcilla A, Mittelbrunn M, Nazarenko I, Nolte-'t Hoen EN, Nyman TA, O'Driscoll L, Olivan M, Oliveira C, Pallinger E, Del Portillo HA, Reventos J, Rigau M, Rohde E, Sammar M, Sanchez-Madrid F, Santarem N, Schallmoser K, Ostenfeld MS, Stoorvogel W, Stukelj R, Van der Grein SG, Vasconcelos MH, Wauben MH, De Wever O. Biological properties of extracellular vesicles and their physiological functions. J Extracell Vesicles. 2015 May 14;4:27066. doi: 10.3402/jev.v4.27066. eCollection 2015. PMID 25979354
- [Background] Fruhbeis C, Helmig S, Tug S, Simon P, Kramer-Albers EM. Physical exercise induces rapid release of small extracellular vesicles into the circulation. J Extracell Vesicles. 2015 Jul 2;4:28239. doi: 10.3402/jev.v4.28239. eCollection 2015. PMID 26142461
- [Background] Sadovska L, Auders J, Keisa L, Romanchikova N, Silamikele L, Kreismane M, Zayakin P, Takahashi S, Kalnina Z, Line A. Exercise-Induced Extracellular Vesicles Delay the Progression of Prostate Cancer. Front Mol Biosci. 2022 Jan 11;8:784080. doi: 10.3389/fmolb.2021.784080. eCollection 2021. PMID 35087866